CLINICAL TRIAL: NCT00878865
Title: Bioequivalence Study Comparing Two Alprazolam 1 mg Tablets; an Open, Randomised, Single Centre, Single Dose Study With Crossover Design in Healthy Subjects
Brief Title: Bioequivalence Study Comparing Two Alprazolam 1 mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: MD, PH.D. Kimmo Ingman, Orion Corporation, Orion Pharma
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0228014
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
Keywords: Alprazolam; bioequivalence
MeSH Terms: interventions — Alprazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alprazolam 1 mg tablet (Experimental): Alprazolam 1 mg tablet
  Interventions: Drug: Alprazolam
- Xanax 1 mg tablet (Active Comparator): Xanax 1 mg tablet
  Interventions: Drug: Alprazolam

INTERVENTIONS:
Drug: Alprazolam — 1 mg tablet one oral dose
  Arms: Alprazolam 1 mg tablet
Drug: Alprazolam — 1 mg tablet
  Other Names: Xanax
  Arms: Xanax 1 mg tablet

SUMMARY:
The objective of the study is to demonstrate the bioequivalence (BE) of two alprazolam 1 mg tablets.

DETAILED DESCRIPTION:
The study is a phase I, open, randomised, crossover, single dose pharmacokinetic study performed in a single centre. The study consists of 2 treatment periods, during which the study subjects will receive the test product and the reference product in a randomised order. During both treatment periods, the study subjects will receive 1 mg of alprazolam as a single oral dose. The study treatments will be administered after an overnight fast (at least 10 h). Blood samples will be drawn during both treatment periods. The planned duration of the study per subject will be 4-5 weeks including a screening visit, 2 treatment periods with a wash-out between the study treatment administrations and a post-treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) obtained
* Good general health ascertained by detailed medical history, and laboratory and physical examinations
* Finnish speaking males and females, 18-55 (inclusive) years of age
* Body mass index > 19 and < 30 kg/m2 (BMI = weight/height2)
* Weight at least 50 kg
* Regular intestinal transit (no recent history of recurrent constipation, diarrhoea, or other intestinal problems).

Exclusion Criteria:

* Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological or psychiatric disease
* Any condition requiring regular concomitant treatment (including vitamins and herbal products) or likely to need any concomitant treatment during the study
* Intake of any medication that could affect the outcome of the study. As an exception, contraceptives intra uterine device (IUD) containing levonorgestrel and hormonal implant are allowed.
* Any clinically significant abnormal laboratory value or physical finding (including electrocardiogram [ECG] and vital signs) that may interfere with the interpretation of test results or cause a health risk for the subject if he/she participates in the study, as judged by the investigator.
* Known hypersensitivity to the active substance(s) or to any of the excipients of the drug
* History of vasovagal collapses
* History of anaphylactic/anaphylactoid reactions
* History of seizures including febrile seizures
* Pregnant or lactating females
* Females of childbearing potential if they are not using proper contraception (IUD, hormonal implant or surgical sterilization, spermicidal foam in conjunction with condom on male partner) (Note: women of childbearing potential with no current sexual relationship can be included without contraception according to the judgement of the investigator).
* Recent or current (suspected) drug abuse or positive result in the drugs abuse test
* Recent or current alcohol abuse (regular drinking more than 21 units per week for males and more than 16 units per week for females [1 unit = 4 cl spirits or equivalent])
* Current use of nicotine containing products more than 5 cigarettes (or equivalent)/day and/or inability to refrain from the use of nicotine containing products during the study (from the screening visit to the end-of-study visit).
* Use of caffeine containing beverages more than 600 mg of caffeine/day and/or inability to refrain from the use of caffeine containing beverages during the treatment periods until 24 h after study treatment administration.
* Blood donation or loss of significant amount of blood within 90 days prior to the first study treatment administration
* Administration of another investigational treatment within 90 days prior to the first study treatment administration
* Unsuitable veins for repeated venipuncture
* Predictable poor compliance or inability to communicate well with the study centre personnel
* Inability to participate in all treatment periods.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Cmax, AUCt and AUC∞ | 48 hours per period

CONTACTS AND LOCATIONS:
Overall Officials: Aila Holopainen, M. Sc., Study Director — Orion Corporation, OrionPharma
Locations (1):
- Orion Pharma phase I unit, Espoo, Finland